CLINICAL TRIAL: NCT01125319
Title: Secondary Adult's Hemophagocytic Lymphohistiocytosis and Innate Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2007/35; 2007-A01109-44 (Registry Identifier: 2007/35)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hemophagocytic Lymphohisticytosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- patients Hemophagocytic lymphohisticytosis group (Other)
  Interventions: Other: blood sample
- group control patient (Other)
  Interventions: Other: blood sample
- healthy control group (Other)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Hemophagocytic lymphohisticytosis (HLH) is a rare and severe disease of genetic origin in children (familial-HLH, F-HLH) or affecting adults secondary to infections, hematologic malignancies or auto-immune diseases (secondary_HLH, S-HLH). F-HLH are due to genetic mutations affecting the genes of perforin or proteins involved in its secretion, resulting in the complete loss of lymphocyte cytotoxicity without affecting lymphocyte number. In S-HLH, the investigators have observed a severe NK cell lymphopenia and a transient loss of cytotoxicity of unknown mechanism. In this study, the investigators will dissect macrophage activation mechanisms as well as NK cytotoxicity inability in adults patients suffering of S-HLH.

Macrophage activation could result from the loss of the retro-control normally exerted by NK cells, thus the investigators will analyze reciprocal interactions of macrophages and NK cells during the acute phase and after recovery of S-HLH.

ELIGIBILITY:
Inclusion Criteria:

Patients Hemophagocytic lymphohisticytosis group:

* Of more than 18 years old
* affected by secondary LH infections with the exception of the HIV, the lymphomes, the néoplasies or the autoimmunes / inflammatory diseases following the criteria of the HLH Society modified in 2004

group control

* Of more than 18 years old
* At the time of the diagnosis either of firstly viral infection (EBV, CMV, parvovirus B19, HSV), is of lymphome cunning(malignant) not - Hodgkinien or of epithelial métastasés cancers, or auto-immune disease (erythemic lupus and disease of Still of the adult only) without associated criteria corresponding to the diagnosis of LHS
* have agreed to benefit from a pregnancy test and from a screening sérologique by the infection by the HIV. These tests that must be negative. In case of positivity of the screening HIV, the patients will be directed to an adequate service.
* Have still received no preliminary treatment for this pathology
* Have agreed to participate in the study and to have signed the form of consent

group healthy control They will have to be unhurt of active infectious pathology, hématologique, auto-immune or neoplastic and have by receipt of immunosuppresseurs treatments during the last 2 years.

Exclusion Criteria:

Patients Hemophagocytic lymphohisticytosis group:

* Minor patients under age 18 or vulnerable (encircled women, private persons of freedom judicially or administratively, adults under guardianship, under guardianship and to express their consent)
* histories of established LHF or episode of LH during the childhood
* patients reached(affected) by infection by the HIV: either histories known for seropositivity and / or of disease, or because of the positivity of the test sérologique realized in the inclusion after consent of the patient.
* Have already benefited from a specific treatment of the LHS

group control

Patients under age 18 and not to belong in one group of vulnerable persons (encircled women, private persons of freedom judicially or administratively, adults under guardianship, under guardianship and to express their consent)

* Patients answering the criteria of diagnosis of LHS
* Patients having already had histories of LH
* Patients having already received the specific treatments of these diseases
* patients reached(affected) by infection by the HIV: either histories known for seropositivity and / or of disease, or because of the positivity of the test sérologique realized in the inclusion after consent of the patient.

group healthy control Patients under age 18 and not to belong in one group of vulnerable persons (encircled women, private persons of freedom judicially or administratively, adults under guardianship, under guardianship and to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the cytotoxicité lymphocytaire | 3 years
  To compare the cytotoxicité lymphocytaire at the patients affected by LHS with regard to 2 groups of subjects controls: a group of patients affected by infections except HIV, by hémopathies or by epithelial métastasés cancers, by autoimmunes / inflammatory pathologies (spread erythemic lupus and disease of Still of the adult) but having no LHS (controls-patients) and a group of healthy subjects.

SECONDARY OUTCOMES:
Study of the mechanisms of the activation macrophagique | 3 years
  Study of the mechanisms of the activation macrophagique

CONTACTS AND LOCATIONS:
Overall Officials: jean robert HARLE, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France